CLINICAL TRIAL: NCT06917261
Title: Evaluation of the Diagnostic Performance of the DM-DIV (in Vitro Diagnostic Medical Device) TestNPass for the Diagnosis of SARS-CoV-2 Infection Using a Nasopharyngeal Sample
Brief Title: Evaluation of the Diagnostic Performance of the TestNPass DM-DIV for SARS-CoV-2 Using a Nasopharyngeal Sample
Acronym: TESTOGRAPH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 38RC24.0309
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: SARS-CoV-2 Infection
Keywords: SARS-CoV-2; Diagnosis; TestNPass; Nasopharyngeal Sample
MeSH Terms: conditions — COVID-19; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cases: 100 cases will be recruited : Patient diagnosed by RT-PCR for a COVID19 (Active Comparator): Diagnostic Test: TestNPass Patients will undergo nasopharyngeal sampling. Grenoble University Hospital lab will perform diagnosis using TestNPass IVDMD. Results won't be used for patient care (only recorded for RESEARCH purpose).
  Interventions: Diagnostic Test: nasopharyngeal swab.
- Controls 300 controls : Patient suspected for a COVID-19 but negative by RT-PCR for a COVID19 (Sham Comparator): Diagnostic Test: TestNPass Patients will undergo nasopharyngeal sampling. Grenoble University Hospital lab will perform diagnosis using TestNPass IVDMD. Results won't be used for patient care (only recorded for RESEARCH purpose).
  Interventions: Diagnostic Test: nasopharyngeal swab.

INTERVENTIONS:
Diagnostic Test: nasopharyngeal swab. — The only additional procedure related to the study is a nasopharyngeal swab.

SUMMARY:
The COVID-19 pandemic has created a major global health crisis that requires a rapid and effective response, particularly in the field of diagnostics.

The first tests used, based on PCR (polymerase chain reaction) performed through a deep nasopharyngeal swab, have shown their limitations in controlling the epidemic. The current need is to develop new tests that are rapid, affordable and easy to use, and that can be used on a large scale in outpatient settings to reduce the burden on healthcare teams. In addition, a test that is easy to produce and can be stored at room temperature would help overcome the significant logistical challenge of regularly testing the general population to specifically isolate carriers of the virus.

In this context, an innovative test called "TestNPass" has been developed. TestNPass is a rapid and affordable antigen test for screening and diagnosis that provides a secure digital passport and/or QR code upon request.

Our aim is to evaluate the diagnostic performance of TestNPass using nasopharyngeal swabs for the detection of SARS-CoV-2 infection.

DETAILED DESCRIPTION:
The COVID-19 pandemic and the global spread of SARS-CoV-2 are historic events in terms of their magnitude and the collective response they have elicited from medical teams, governments and the general public. This situation requires a rapid and effective response to find solutions, particularly in the field of diagnostics.

While the initial tests used were based on PCR (polymerase chain reaction) and deep nasopharyngeal swabs, this approach has shown its limitations in controlling the epidemic. The significant logistical resources required for its implementation limit its large-scale use beyond what is currently being done. In addition, deep nasopharyngeal sampling is not feasible for repeated testing of healthy populations as part of primary screening.

The current need is to develop new point-of-care (PoC) testing methods that are rapid, affordable and easy to use. These characteristics would allow mass use in outpatient settings, reducing the burden on healthcare teams. In addition, a test that is easy to produce and can be stored at room temperature would address the immense logistical challenge of regularly testing the general population to specifically isolate virus carriers.

In this context, an innovative test called "TestNPass" has been developed by the Grenoble-based start-up company Grapheal. TestNPass is a rapid and low-cost antigen test for screening and diagnosis that delivers a secure digital passport and/or QR code on request. This type of device could also be used to detect various antigens, such as those of influenza, streptococcus A or shingles.

Our objective in this study is to evaluate the diagnostic performance of an in vitro diagnostic medical device (IVD) for the detection of SARS-CoV-2 infection using a nasopharyngeal swab. To achieve this, we will take an additional nasopharyngeal swab sample immediately after the sample taken as part of routine health care.

A total of 400 adult participants who require a nasopharyngeal swab for their medical care will be enrolled in this study. The only additional procedure involved in the study is the collection of a second nasopharyngeal swab. The study consists of a single visit (1 day).

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age
* Consulting or hospitalized at the University Hospital of Grenoble Alpes, for whom a SARS-CoV-2 RT-PCR test via nasal swab is considered due to symptoms or context (hospitalization in a double room, ongoing epidemic outbreak)
* Having provided informed consent to participate in the study.
* Patient having the rights to French social insurance

Exclusion Criteria:

* Contraindication to nasopharyngeal swabbing:
* Anatomical abnormalities or medical conditions:
* Severe nasal septum deviation or nasal polyps
* History of recent nasal or facial surgery
* Severe sinusitis or nasal infections
* Bleeding disorders
* Extreme sensitivity or phobias related to medical procedures
* Participation in an exclusion period of another SARS-CoV-2 performance study: Minors

Pregnant or breastfeeding women, Individuals under guardianship or curatorship, Individuals deprived of liberty or involuntarily hospitalized, Individuals under administrative or judicial supervision, Persons unable to provide informed consent

* Staff with a hierarchical relationship with the principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Analytics performance (specificity) of TestNPass | DAY0 (single visit study, day of COVID19 diagnosis)
  Specificity in % of TestNPass using a nasopharyngeal swab. The specificity target is set at 99%.

SECONDARY OUTCOMES:
Analytics performance (Sensitivity) of TestNPass | DAY0 (single visit study, day of COVID19 diagnosis)
  Sensitivity in %, positive predictive value (PPV), negative predictive value (NPV), positive likelihood ratio (PLR), and negative likelihood ratio (NLR).

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - University Hospital of Grenoble, emergency department, Grenoble
  - University Hospital of Grenoble, infectious disease department, Grenoble

IPD SHARING:
Plan to Share IPD: Undecided